CLINICAL TRIAL: NCT06010368
Title: The Effect of Intramyometrial Tranexamic Acid Versus Intramyometrial Oxytocin in Reducing Blood Loss During and After Elective Cesarean Section in Term Primigravida: A Double-blinded, Randomized, Comparative-placebo Trial
Brief Title: Comparing Intramyometrial Tranexamic Acid and Oxytocin for Blood Loss in Cesarean Section
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed nagy shaker ramadan, Assistant lecturer of obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AN2023-3
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Cesarean Section Complications; Tranexamic Acid; Oxytocin; Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid; Oxytocin

STUDY DESIGN:
Intervention Model Description: patients assigned to the oxytocin group (n = 75): 5 I.U of oxytocin (syntocinone 5 I.U/1ML NONARTIS-EGYPT) shall be watered down in 10 cc of saline, and 5 cc shall be injected into each uterine corn before the placental separation. In TXA group (n=75): 1 g from tranexamic acid (kapron®, Amoun, Egypt) shall also be watered down in 10 cc of Saline, and 5 cc shall be injected in each uterine corn before the placenta is separated.
Who Masked: Participant, Outcomes Assessor
Masking Description: A double-blind study is one in which neither the participants nor the experimenters know who is receiving a particular treatment. This procedure is utilized to prevent bias in research results. Double-blind studies are particularly useful for preventing bias due to demand characteristics or the placebo effect. In a double-blind study, the investigators who interact with the participants would not know who will receive the actual drug and who will receive a placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Tranexamic acid group (Experimental): In TXA group (n=75): 1 g from tranexamic acid (kapron®, Amoun, Egypt) shall also be watered down in 10 cc of Saline, and 5 cc shall be injected in each uterine corn before the placenta is separated.
  Interventions: Drug: Tranexamic acid injection
- Group 2: oxytocin group (Experimental): to the oxytocin group (n = 75): 5 I.U of oxytocin (syntocinone 5 I.U/1ML NONARTIS-EGYPT) shall be watered down in 10 cc of saline, and 5 cc shall be injected into each uterine corn before the placental separation
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Tranexamic acid injection — In TXA group (n=75): 1 g from tranexamic acid (kapron®, Amoun, Egypt) shall also be watered down in 10 cc of Saline, and 5 cc shall be injected in each uterine corn before the placenta is separated.
  Other Names: kapron
  Arms: Group 1: Tranexamic acid group
Drug: Oxytocin — the oxytocin group (n = 75): 5 I.U of oxytocin (syntocinone 5 I.U/1ML NONARTIS-EGYPT) shall be watered down in 10 cc of saline, and 5 cc shall be injected into each uterine corn before the placental separation
  Other Names: syntocinone
  Arms: Group 2: oxytocin group

SUMMARY:
Cesarean section is the most prevalent operation among women globally, 10-15% (1, 2). Recent research has shown Egypt to be the third-largest country globally, with an estimated 52% cesarean sections (3). However, the cesarean section has many serious complications, including the primary postpartum hemorrhage (PPH) (4). During labor, the average blood loss is about 300 to 400 ml. Bleeding postpartum is known as losing over five hundred milliliter of blood following a vaginal birth and losing over one thousand milliliter after the cesarean section (5). The prime cause of maternal death rate is postpartum bleeding, predominately in poor countries, and the estimated mortality number due to postpartum bleeding is one hundred thousand per year (6). Therefore, it is essential to reduce bleeding during and after CS to diminish maternal mortality and morbidity (7). The most successful technique for decreasing PPH is the active third stage labor management, requiring prophylactic uterotonic drugs like oxytocin, ergometrine malate, prostaglandins (E1, E2, and F2α), and combinations of them, or hemostatic agent as tranexamic acid (Kapron) and Etamsylate (Dicynon) (8, 9).

DETAILED DESCRIPTION:
Study design: This study is a double-blinded prospective randomized comparative Clinical trial to compare and evaluate the effectiveness of intra-myometrial oxytocin injection and intra-myometrial tranexamic acid injection in reducing the risk of postpartum bleeding after cesarean delivery in primigravida at term. The study will be conducted in Maternity hospital, Fayoum University, Fayoum, Egypt, during june 2024 to December 2025. After The Ethical Research Committee approval on study protocol, fifty primigravida women at term pregnancy, undergoing elective cesarean delivery will be divided and allocated randomly into two groups after fulfillment eligibility criteria. Fifty women will be included in this clinical study at admission to the labor ward. Written informed permission will be acquired following advising about this study and potential implications. A history in details and clinical examination for all patients to rule out general health problems. Vaginal and Abdominal examinations will be done. Routine preoperative investigations and obstetric ultrasound examinations will be done for all women to ensure that all inclusion criteria were present. The computer will be used for randomization to allocate the patients into two equal groups. Randomization cards will be produced, sealed and stored; sequentially black wrappers will be numbered. The hospital pharmacy is producing packages, and physicians and nurses were unaware of their contents. For the entire length of the trial, all study personnel and participants are blinded to therapy. A senior registrar will execute a cesarean section before the commencement of research, which performs at least 300 cesarean sections. All cesarean section will be operated via spinal anesthesia; the abdomen will be entered through the Pfannenstiel incision. The sealed envelope is carried to the operating room and transferred without informing the researcher or the patients about their contents. The anesthesiologist is administering the medication (Oxytocin or tranexamic acid). After fetal birth and before placental delivery, patients assigned to the oxytocin group (n = 75): 5 I.U of oxytocin (syntocinone 5 I.U/1ML NONARTIS-EGYPT) shall be watered down in 10 cc of saline, and 5 cc shall be injected into each uterine corn before the placental separation. In TXA group (n=75): 1 g from tranexamic acid (kapron®, Amoun, Egypt) shall also be watered down in 10 cc of Saline, and 5 cc shall be injected in each uterine corn before the placenta is separated. The primary outcome is to decrease Intra and postoperative blood loss to reduce PPH risk after CS. After a skin incision, the estimated blood loss would begin. The towels are weighted in (mg) with their covers, using an exact digital balance, before and following the operation, and the weight variation is measured between dryish and saturated towels. Blood loss is counted as follows during the operation: volume contents in the suction container in (ml) (X), the towel weight variation in (gm), (Y) (weight of saturated towels in (gm) - weight of dry towel in (gm)), the amniotic liquid amount in (ml) (Z). Operational blood loss in (ml) = (X+Y) - Z (18). All women are calculated according to the underlying law for permissible blood loss. Allowable blood loss = The estimated volume of blood x (initial hematocrit - final lowest acceptable hematocrit)/ initial hematocrit, an estimated volume of blood = weight of the patient in (kg) multiplies by average volume of blood (75-85 ml/kg) (19).

ELIGIBILITY:
nclusion Criteria:

* Women booked for a primary elective cesarean section, not in active labor
* Aged between 20-40 years.
* BMI 18.5-29.9 kg/ m2 pre-pregnancy weight
* Term pregnancies (Early term: between 37 weeks, 0 days and 38 weeks, 6 days. Full term: between 39 weeks, 0 days and 40 weeks, 6 days. Late term: between 41 weeks, 0 days and 41 weeks, 6 days).
* Singleton pregnancies.
* Indication of elective cesarean section (Malpresentation, Malposition, Cephalopelvic disproportion, active herpes)
* Fetal macrosomia (Macrosomia is defined as birth-weight over 4,000 g irrespective of gestational age)
* Certain congenital fetal malformation and skeletal disorders (Several congenital anomalies are controversial indications for cesarean delivery; these include fetal neural tube defects (to avoid sac rupture), particularly defects that are larger than 5-6 cm in diameter as anterior cystic hygroma vascular sacrococcygeal teratoma, giant omphalocele and hydrocephalus with an enlarged biparietal diameter, and some skeletal dysplasia such as type III osteogenesis imperfecta. (Hamrick et al., 2008)

Exclusion Criteria:

* Placenta previa.
* Maternal hypertension and Preeclampsia.
* Diabetes mellitus.
* Severe medical disorder (renal or hepatic).
* Multiple Fibroid uterus.
* Multiple pregnancies.
* Polyhydramnios.
* Previous uterine surgery as myomectomy.
* Contraindication to spinal anesthesia.
* Blood coagulopathy and bleeding disorder.
* Marked maternal anemia (Preoperative hemoglobin <9 gm/dl).
* Contraindications to TXA or oxytocin therapy (e.g. allergy)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Blood loss | 24 hours
  Estimation of Intraoperative and postoperative blood loss.

SECONDARY OUTCOMES:
Need of extra utero-tonic drugs | 2 hours
  Need of extra utero-tonic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed N Afifi, MD, Principal Investigator — Kafrelsheikh University; Ahmed N Shaker, MD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Suez Canal University, Ismailia, Egypt

REFERENCES:
- [Background] El-Zanati FJICAfPM, Economic SRib, Knowledge SJU, B PoH. Egypt Health Issues Survey, Ministry of Health and Population, El-Zanaty and Associates and, ICF International. 2015:25-50.
- [Background] Kebede BA, Abdo RA, Anshebo AA, Gebremariam BM. Prevalence and predictors of primary postpartum hemorrhage: An implication for designing effective intervention at selected hospitals, Southern Ethiopia. PLoS One. 2019 Oct 31;14(10):e0224579. doi: 10.1371/journal.pone.0224579. eCollection 2019. PMID 31671143
- [Background] Brun R, Spoerri E, Schaffer L, Zimmermann R, Haslinger C. Induction of labor and postpartum blood loss. BMC Pregnancy Childbirth. 2019 Jul 25;19(1):265. doi: 10.1186/s12884-019-2410-8. PMID 31345178
- [Result] Visconti F, Quaresima P, Rania E, Palumbo AR, Micieli M, Zullo F, Venturella R, Di Carlo C. Difficult caesarean section: A literature review. Eur J Obstet Gynecol Reprod Biol. 2020 Mar;246:72-78. doi: 10.1016/j.ejogrb.2019.12.026. Epub 2020 Jan 7. PMID 31962259
- [Result] Boerma T, Ronsmans C, Melesse DY, Barros AJD, Barros FC, Juan L, Moller AB, Say L, Hosseinpoor AR, Yi M, de Lyra Rabello Neto D, Temmerman M. Global epidemiology of use of and disparities in caesarean sections. Lancet. 2018 Oct 13;392(10155):1341-1348. doi: 10.1016/S0140-6736(18)31928-7. PMID 30322584